CLINICAL TRIAL: NCT03235141
Title: Local Pharmacokinetics of Azithromycin Eye Drops in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Zhuhai Essex Bio-Pharmaceutical Company Limited (Unknown); Panacea Technologies (Other)
Responsible Party: Principal Investigator, Xiuli Zhao, Director of Phase I Clinical Trial Center, Beijing Tongren Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ESSEX-AOS-PK-2001
Record Dates: First submitted 2017-07-05; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Bacterial Conjunctivitis
Keywords: Azithromycin eye drops; Local Pharmacokinetics
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: There are 8 subjects will be enrolled in pre-test, each subject was sampled in two eyes and each subject participated in two cycles of the trial. 8 subjects, 16 eyes participated in the study, 32 samples of tears total .
  There are 48 subjects will divided into group A and group B randomly . subjects of Group A will given the first test drug, elution after the control drug; Subjects of Group B will given the first control drug, elution given to the test drug.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- azithromycin eye drops by essex (Experimental): In one cycle, give the azithromycin eye drops by essex,2.5ml/25mg，1 drop，once. In the second cycle(after 14 days elution）,give the AzaSite eye drops,2.5ml/25mg，1 drop，once.
  Interventions: Drug: azithromycin eye drops by essex; Drug: azithromycin eye drops
- AzaSite (Active Comparator): In one cycle, give the AzaSite eye drops,2.5ml/25mg，1 drop，once. In the second cycle(after 14 days elution）,give the azithromycin eye drops by essex,2.5ml/25mg，1 drop，once.
  Interventions: Drug: azithromycin eye drops by essex; Drug: azithromycin eye drops

INTERVENTIONS:
Drug: azithromycin eye drops by essex — azithromycin eye drops,2.5ml/25mg,by ZHUHAI ESSEX BIO-PHARMACEUTICAL),
Drug: azithromycin eye drops — azithromycin eye drops,2.5ml/25mg ,by Oak Pharmaceuticals, Inc subsidiary of Akorn, Inc
  Other Names: AzaSite

SUMMARY:
To compare the pharmacokinetic behavior of azithromycin eye drops in the tear with the original azithromycin eye drops, and evaluate the release behavior of both in the eye.

DETAILED DESCRIPTION:
There are 48 patients will divided into group A and group B randomly . subjects of Group A will given the first test drug, elution after the control drug; Subjects of Group B will given the first control drug, elution given to the test drug.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old, male or female;
* BMI in the range of 19 to 28;
* eyes corrected visual acuity should be ≥ 1.0, intraocular pressure, slit lamp and fundus examination were normal, tear secretion function is normal;
* Good compliance and voluntarily signed consent.

Exclusion Criteria:

* Have eye disease or systemic disease;
* physical examination, laboratory tests, ECG and chest X-ray examination abnormalities and has clinical significance;
* HBsAg, anti-HCV and HIV positive;
* those who used eye drops two weeks before the test and who used any dosage form of azithromycin;
* known to azithromycin or macrolide-related varieties of allergies or serious adverse reactions;
* need to wear contact lenses during the test;
* history of internal surgery or laser surgery history;
* participated in other drug clinical trials in the past three months;
* pregnant women and lactating women, or in the growth period without taking effective contraceptive measures, menstrual period women;
* mental illness or alcohol, history of drug abuse or inability to collaborate;
* Any other circumstances that the investigators consider are unfit to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | The tear samples were taken at 8 time points after administration,10 minutes,half hour,2 hours,4 hours,8 hours,12 hours,24 hours,36 hours
  The tear samples were taken at 8 time points after administration,10 minutes,half hour,2 hours,4 hours,8 hours,12 hours,24 hours,36 hours，The AUC of the test drug and the control drug was calculated at the average concentration of each point

SECONDARY OUTCOMES:
Cmax | The tear samples were taken at 8 time points after administration,10 minutes,half hour,2 hours,4 hours,8 hours,12 hours,24 hours,36 hours
  The tear samples were taken at 8 time points after administration,10 minutes,half hour,2 hours,4 hours,8 hours,12 hours,24 hours,36 hours，The Cmax of the test drug and the control drug was calculated at the average concentration of each point
AE | from the ICF signed to the end of the trial,through study completion, an average of 1 year
  compared the laboratory test values before and after treatment,according to the study drug use, calculate the number of cases, the number of cases and the incidence of adverse reactions.
SAE | from the ICF signed to the end of the trial,through study completion, an average of 1 year
  Any serious adverse events that occur during the clinical study, whether or not related to the drug should be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No